CLINICAL TRIAL: NCT00261248
Title: Phase 2 Clinical Trial of Vaginal Mucosal Immunization for Recurrent Urinary Tract Infections
Brief Title: Vaccine for Recurrent Urinary Tract Infections in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1996-295; DK-30808
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2003-09

CONDITIONS: Recurrent Urinary Tract Infections in Women
Keywords: Phase 2; Vaccine; Urinary Tract Infection; Vaginal Mucosal
MeSH Terms: conditions — Urinary Tract Infections | interventions — Immunization

INTERVENTIONS:
Biological: Immunization with inactivated bacteria

SUMMARY:
The purpose of this study is determine whether a vaginal mucosal vaccine given to women with a history of recurrent urinary tract infections can reduce the number of infections occurring in a six-month study period, as compared to placebo treatment.

DETAILED DESCRIPTION:
Recurrent urinary tract infections (UTIs) affect approximately 10% of women in the United States. Since antibiotic prophylaxis is not always effective, alternate treatments need to be developed. One such treatment would be immunization with a vaccine containing bacteria known to cause these infections. The objective of the study is to immunize susceptible women with inactivated bacteria contained in a vaginal suppository and to monitor the rates of reinfection compared to a group of women treated with placebo suppositories. Each group of patients will receive a total of six suppositories in the first four-months of the six-month study during which all UTIs and side effects will be recorded. The infection rates between vaccine- and placebo-treated women will be statistically analyzed to determine vaccine efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Three or more urinary tract infections in the previous year

Exclusion Criteria:

* Neurogenic bladder
* Interstitial cystitis
* Urinary diversion
* Kidney stones
* Indwelling catheter

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 1996-11; Study Completion 2003-12

PRIMARY OUTCOMES:
Rate of re-infection over the study

SECONDARY OUTCOMES:
Infection-free status at completion of study

CONTACTS AND LOCATIONS:
Overall Officials: David T Uehling, M.D., Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- [Background] Uehling DT, Hopkins WJ, Beierle LM, Kryger JV, Heisey DM. Vaginal mucosal immunization for recurrent urinary tract infection: extended phase II clinical trial. J Infect Dis. 2001 Mar 1;183 Suppl 1:S81-3. doi: 10.1086/318839. No abstract available. PMID 11171022